CLINICAL TRIAL: NCT06549179
Title: Validation Study of the Screening Performance of the French Version of the Autism Mental Status Examination Scale as a Tool for Identifying Autism Spectrum Disorder in Adults
Brief Title: Validation Study of the Performance of the French Version of the Autism Mental Status Examination Scale as a Tool for Identifying Autism Spectrum Disorder in Adults
Acronym: AUTI-SCREEN
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210995
Record Dates: First submitted 2024-02-14; First posted 2024-08-12 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Mental Status Disorder; Adult
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients evaluated by AMSE: Adult patients seeking ASD diagnostic evaluation in an expert center.
  Interventions: Diagnostic Test: AMSE

INTERVENTIONS:
Diagnostic Test: AMSE — Evaluation of the performance of the French-language AMSE tool used by non-expert psychiatrists and psychologists, trained in the tool, in the identification of ASD in adults.

SUMMARY:
To improve diagnosis of Autism Spectrum Disorder (ASD), expert centers have been set up in France since 2000/2010. However, waiting times in these centers are long, mean of 19 months for adults, and more than half the people seen do not end up with an ASD, even though referral by a psychiatrist is increasingly required.

Therefore, validated diagnostic tools for screening before referral are needed. The Autism Mental Status Exam (AMSE), a 8-item tool, which is quick and easy to use, appears to have excellent sensitivity (0.91) and specificity (0.93). However, this tool was only evaluated when used by experts and on a sample of 50 patients.

The hypothesis of this study is that the AMSE, used by non-expert psychiatrists, has sufficiently good diagnostic performance (minimal sensitivity and specificity of respectively 93% and 65%) to be used in screening adults with suspected ASD.

DETAILED DESCRIPTION:
Patients who contact one of the expert centers participating in the study for an ASD diagnostic evaluation are first referred, as in usual care, to a non-expert psychiatrist or psychologist (from a list of professionals provided by the center and previously trained to the AMSE) to complete a pre-evaluation file. For the study the AMSE and a brief AMSE-filling guide is added to the file.

Seven days to 12 months after, patients have a 2-day (consecutive or separated by a maximum of 2 months) full ASD evaluation in the expert center with a final diagnosis made by the expert multidisciplinary team according to Diagnostic and Statistical Manual (DSM)-5 criteria for ASD.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years of age or older
* Patient who has requested, either personally, through a relative, or through a healthcare professional, a diagnostic evaluation at a center specializing in ASD diagnosis.
* Patient covered by national health insurance

Exclusion Criteria:

* Patient who has previously undergone a diagnostic assessment resulting in a diagnosis of Autism Spectrum Disorder (ASD) made by a psychiatrist or child psychiatrist
* Absence of informed consent (patient or his/her legal guardian)
* Pregnant or breast-feeding
* Patient deprived of freedom
* Non-French-speaking patient and/or parents and/or legal guardians
* AMSE not, incorrectly or inadequately completed by non-expert psychiatrist or psychologist
* Patient covered by Aide Medicale d'Etat (AME)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adults (aged 18 or over) requesting a diagnostic assessment in an expert center.
Sampling Method: Non-Probability Sample
Enrollment: 410 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of the AMSE tool rated by a non-expert psychiatrist or psychologist but trained to in ASD diagnosis and to the tool, and considered here as the index test, in identifying ASD in adults. | 0-12 months from AMSE rating
  Diagnostic performance as measured by sensitivity, specificity, area under the receiver operating characteristic curve for different thresholds, compared to the reference standard.
  The reference standard is the final diagnosis made by the expert multidisciplinary team according to DSM-5 criteria for ASD, based on all routine assessments, i.e.: anamnesis and use of standardized tools with, at best, Autism Diagnostic Observation Scale (ADOS-2) (if fluid language) and Autism Diagnostic Interview (ADI-R) (if accompanying parent present), or, alternatively : Adult Asperger Assessment (AAA), (ASD-DA), Echelle des Comportements Répétés et Restreints (EC2R), Pervasive Developmental Disorder in Mental Retardation Scale (PDD-MRS).

SECONDARY OUTCOMES:
Other accuracy measures of the AMSE tool rated by a non-expert psychiatrist or psychologist trained to the tool, in identifying ASD in adults. | 0-12 months from AMSE rating
  Positive and negative likelihood ratio, positive and negative predictive values for different thresholds, compared to the reference standard.
Accuracy of the AMSE tool rated by a non-expert psychiatrist or psychologist trained to the tool, in identifying ASD in adults, according to the presence or absence of an intellectual disability (Intellectual coefficient<70 measured on the WAIS-IV). | 0-12 months from AMSE rating
  Diagnostic performance as measured by sensitivity, specificity, positive and negative likelihood ratio, positive and negative predictive values, area under the receiver operating characteristic curve for different thresholds, compared to the reference standard.
Accuracy of the AMSE tool, rated by an expert psychiatrist or psychologist, in identifying ASD in adults. | 0-12 months from AMSE expert rating
  Diagnostic performance as measured by sensitivity, specificity, positive and negative likelihood ratio, positive and negative predictive values, area under the receiver operating characteristic curve for different thresholds, compared to the reference standard.
Differential diagnoses | 0-12 months from AMSE rating
  Presence and nature of differential diagnosis (personality disorders, anxiety disorders, schizophrenia spectrum disorders, other neurodevelopmental disorders) made by the expert multidisciplinary team.
AMSE score according to differential diagnosis | 0-12 months from AMSE rating
  Mean, standard deviation, median, min, max, inter quartile range of AMSE rated by a non-expert psychiatrist or psychologist trained to the tool
Acceptability on the AMSE tool by non-expert psychiatrists or psychologists trained to use the tool. | Immediately after AMSE rating
  Perception of the tool's relevance, ease of completion, completion time (duration in minutes), use of written guide, use of self-training video tutorial, and previous experience with the tool.
Feedback on the AMSE tool by non-expert psychiatrists or psychologists trained to use the tool. | Immediately after AMSE rating
  Perception of the tool's relevance, ease of completion, completion time (duration in minutes), use of written guide, use of self-training video tutorial, and previous experience with the tool.
Exploratory : predictive model of ASD diagnosis | 0-12 months from AMSE rating
  Predictive model of ASD diagnosis for patient with intellectual disability, with AMSE tool rated by a non-expert psychiatrist or psychologist trained to the tool.
Exploratory : predictive model of ASD diagnosis | 0-12 months from AMSE rating
  Predictive model of ASD diagnosis for patient without intellectual disability, with AMSE tool rated by a non-expert psychiatrist or psychologist trained to the tool.

CONTACTS AND LOCATIONS:
Locations (1):
- Pitié-Salpêtrière Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients. Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor.
Access Criteria: Researchers who provide a methodologically sound proposal.